CLINICAL TRIAL: NCT00750633
Title: A Phase III Study of an Otic Formulation in Acute Otitis Externa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-07-13
Record Dates: First submitted 2008-09-08; First posted 2008-09-10 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Acute Otitis Externa
Keywords: swimmer's ear; ear drops; ear infection; ear pain; ear inflammation
MeSH Terms: conditions — Otitis Externa; Otitis; Earache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Moxidex (Experimental): Moxidex otic solution
  Interventions: Drug: Moxidex otic solution; Device: Tympanostomy tubes
- Moxifloxacin (Active Comparator): Moxifloxacin otic solution
  Interventions: Drug: Moxifloxacin otic solution; Device: Tympanostomy tubes
- Dexamethasone (Active Comparator): Dexamethasone phosphate otic solution
  Interventions: Drug: Dexamethasone phosphate otic solution; Device: Tympanostomy tubes

INTERVENTIONS:
Drug: Moxidex otic solution — 4 drops in the infected ear(s) twice daily (morning and evening) for 7 days
  Arms: Moxidex
Drug: Moxifloxacin otic solution — 4 drops in the infected ear(s) twice daily (morning and evening) for 7 days
  Arms: Moxifloxacin
Drug: Dexamethasone phosphate otic solution — 4 drops in the infected ear(s) twice daily (morning and evening) for 7 days
  Arms: Dexamethasone
Device: Tympanostomy tubes — Tubes surgically inserted through the ear drum for the treatment of recurrent otitis media with effusion in children

SUMMARY:
The purpose of this study is to determine if an otic formulation is safe and effective for the treatment of acute otitis externa (AOE).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AOE based on clinical observation and of presumed bacterial origin
* A minimum combined score of ≥4 in at least 1 affected ear at the Day 1 exam for tenderness, erythema, and edema
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Duration of pretherapy signs or symptoms of AOE greater than four (4) weeks
* Presence of a tympanostomy tube or perforated tympanic membrane in the treated ear(s). Patients with a history of tympanic membrane perforation should not be enrolled unless the absence of a current perforation can be confirmed at Visit 1 prior to enrollment
* Clinically diagnosed chronic suppurative otitis media, acute otitis media, acute otorrhea in patients with tympanostomy tubes, or malignant otitis externa
* Known or suspected ear infection of fungal or mycobacterial origin
* Prior otologic surgery within 6 months of study entry
* Seborrheic dermatitis or other skin conditions of the external auditory canal
* Current or prior history of an immunosuppressive disorder (e.g., HIV positive) or current immunosuppressive therapy (e.g., cancer chemotherapy) or known acute or chronic renal disorders or active hepatitis
* Diabetic patients (controlled or uncontrolled) based upon assessment by Investigator
* Any systemic disease or disorder, complicating factor or structural abnormality that would negatively affect the conduct or outcome of the study [e.g., cleft palate (including repairs), Downs Syndrome, and cranial facial reconstruction]
* Any current known or suspected infection (other than AOE) requiring systemic antimicrobial therapy
* Use of prohibited medications or inadequate washout of any medication listed in protocol
* Concomitant use of topical or oral analgesics (i.e., NSAIDs and aspirin products) which may have anti inflammatory effects. Patients on low dose aspirin therapy (81 mg per day) at the time of enrollment may be enrolled and continue the low dose aspirin during the study. Use of acetaminophen ("Tylenol") is permitted during the trial
* Other protocol-defined exclusion criteria may apply

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Clinical Cure | Day 3
Clinical Cure | Day 12

SECONDARY OUTCOMES:
Microbiological Success | Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Contact Alcon Call Center, Study Director — 1-888-451-3937